CLINICAL TRIAL: NCT03328000
Title: Radiological Re-evaluation of Failed Anastomotic Uretheroplasty for PFUDDI Using Computed Tomographic Urethrography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Aliaboeihayagan Ali Mohammed, resident doctor, Assiut University
Other Study IDs: failed urethroplasty
Record Dates: First submitted 2017-10-01; First posted 2017-11-01 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Failed Anastomotic Urethroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CTU and MR urethrography — computed tomographic and Magnetic Resonance Urethrography.

SUMMARY:
Estate vlue of CTU in evaluation of failed anastomotic urethroplasty for pelvic fracture urethral distraction defect injury [PFUDDI] combared to retrograde urethrography and voiding cysto-urethrography .

DETAILED DESCRIPTION:
Blunt pelvic trauma results in posterior urethral distraction defects (PUDDs) in ª10% of cases; such injury commonly involves the membranous urethra at the point of departure from the bulbospongiosum, at the prostatomembranous junction, or at any point between its departure and the apex of the prostate [1]. PUDDs are complex pathologically, involving displacement and misalignment of the severed urethral ends with intervening and surrounding ﬁbrosis. Detached bony fragments and callus formation add to the pathological complexity. For a successful repair of a PUDD it is necessary to identify the speciﬁc anatomy of the distraction defect before undertaking any treatment[2].

Currently most PFUDDI are associated with trauma as an etiology. Posterior urethral disruption occurs in 4-14% of pelvic ring fractures and 80-90% of posterior urethral injuries are associated with pelvic fractures[4]. Sixty-five percent of post-traumatic posterior urethral injuries are complete[5]. Following trauma the ruptured urethra is usually replaced by fibrosis and in between there is no lumen. Anastomotic urethroplasty is a well established procedure to deal with posterior urethral strictures and gives very good long-term results[6,7].

The success rate of repeat surgery for failed urethroplasty is reported to be less than that for primary urethroplasty. Jakse et al;reported a 71% failure rate following end-to-end urethroplasty with a history of prior urethroplasty[8].

The success rate of end-to-end anastomosis varies from 77 to 95% as described by different series[9,10,11,12]There are very few reports regarding urethroplasty for previously failed PFUDDI[13,14],The most common causes of failure of urethroplasty are the inadequate excision of the strictured segment and surrounding fibrosis, improper case selection and ischemia[14].

For a successful repair of a PFUDDI it is necessary to identify the specific anatomy of the distraction defect before undertaking any treatment, The classic approach for evaluating a PFUDDI is through Retrograde Urethrography [RUG] and Voiding cysto-urethrography (VCUG), particularly while the patient is attempting to void. However, this study can often give a false interpretation of the exact anatomy of the distraction defect on many occasions[15].

It often cannot provide an accurate determination of the defect length because of poor prostatic urethral filling and it provides little information on the extent of corpus spongiosal fibrosis or prostatic displacement[15].

CTCUG was more informative than conventional radiology in several aspects; the location and the length of the distraction defect; the direction of alignment or misalignment; the bone anatomy (ectopic fragments, callus); and the presence of additional urinary pathology (ﬁstulae, false passages, diverticulae)[2].

ELIGIBILITY:
Inclusion Criteria:

* 1-patient with normal bladder. 2-Patient with fructure pelvis.

Exclusion Criteria:

* 1-Patient without fracture pelvis. 2-Patient with other pathology as neurogenic bladder.

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: patients with failed anastomotic uretheroplasty for PFUDDI.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of failed anastomotic urethroplasty for pelvic fracture urethral distraction defect injury[PFUDDI], Measurement of the actual length and location of the defect.and detection of bony abnormality as fragment affecting the healing process. | 2years
  Patient with failed anastmotic urethroplasty will undergo CTU to show if they will provide more data about the anatomy of the defect including lenth degree of the fibrosis pelvic blood supply and presence of bone defect affecting healing or any other finding can not be evaluated by other diagnostic measures.